CLINICAL TRIAL: NCT01262391
Title: A Multicenter, Open-label, Single Ascending Dose Study to Evaluate Pharmacokinetics, Safety and Tolerability of Solifenacin Succinate Suspension in Pediatric Patients Aged 5 to 17 Years (Inclusive) With Overactive Bladder (OAB)
Brief Title: Single-dose Study to Assess Pharmacokinetics of Solifenacin Succinate Suspension in Children and Adolescents
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 905-CL-075; 2009-017197-21 (EudraCT Number)
Record Dates: First submitted 2010-11-01; First posted 2010-12-17 (Estimated); Last update posted 2024-10-22 (Actual); Status verified 2024-10

CONDITIONS: Urinary Bladder, Overactive
Keywords: Overactive bladder; Solifenacin suspension; Pharmacokinetics; Single-dose; Pediatric
MeSH Terms: conditions — Urinary Bladder, Overactive | interventions — Solifenacin Succinate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- AD-PED 2.5 mg (Experimental): Male and female adolescents aged 12 to less than 18 years old who receive pediatric equivalent dose (PED) of 2.5 mg of solifenacin succinate.
  Interventions: Drug: Solifenacin succinate suspension 2.5 mg
- AD-PED 5 mg (Experimental): Male and female adolescents aged 12 to less than 18 years old who receive PED of 5 mg of solifenacin succinate.
  Interventions: Drug: Solifenacin succinate suspension 5 mg
- AD-PED 10 mg (Experimental): Male and female adolescents aged 12 to less than 18 years old who receive PED of 10 mg of solifenacin succinate.
  Interventions: Drug: Solifenacin succinate suspension 10 mg
- CH-PED 2.5 mg (Experimental): Male and female children aged 5 to less than 12 years old who receive PED of 2.5 mg of solifenacin succinate.
  Interventions: Drug: Solifenacin succinate suspension 2.5 mg
- CH-PED 5 mg (Experimental): Male and female children aged 5 to less than 12 years old who receive PED of 5 mg of solifenacin succinate.
  Interventions: Drug: Solifenacin succinate suspension 5 mg
- CH-PED 10 mg (Experimental): Male and female children aged 5 to less than 12 years old who receive PED of 10 mg of solifenacin succinate.
  Interventions: Drug: Solifenacin succinate suspension 10 mg

INTERVENTIONS:
Drug: Solifenacin succinate suspension 2.5 mg — Adolescents and children are given a single dose of solifenacin succinate liquid suspension orally via syringe in the morning of day 1 followed by a glass of water. Doses are calculated per weight of the participant, targeting to have equivalent doses of 2.5 mg of solifenacin once daily in adults.
  Other Names: YM905
  Arms: AD-PED 2.5 mg; CH-PED 2.5 mg
Drug: Solifenacin succinate suspension 5 mg — Adolescents and children are given a single dose of solifenacin succinate liquid suspension orally via syringe in the morning of day 1 followed by a glass of water. Doses are calculated per weight of the participant, targeting to have equivalent doses of 5 mg dose of solifenacin once daily in adults.
  Other Names: YM905
  Arms: AD-PED 5 mg; CH-PED 5 mg
Drug: Solifenacin succinate suspension 10 mg — Adolescents and children are given a single dose of solifenacin succinate liquid suspension orally via syringe in the morning of day 1 followed by a glass of water. Doses are calculated per weight of the participant, targeting to have equivalent doses 10 mg dose of solifenacin once daily in adults.
  Other Names: YM905
  Arms: AD-PED 10 mg; CH-PED 10 mg

SUMMARY:
This single-dose study will investigate how well solifenacin suspension is taken up, how long it stays in the body and how well it will be tolerated in children and adolescents aged 5-17 years with symptoms of overactive bladder.

DETAILED DESCRIPTION:
This is a multicenter, open-label, sequential, single ascending dose study. The study will consist of three treatment groups in children and three treatment groups in adolescents, targeting equivalent exposure to the 2.5, 5 and 10 mg doses o.d. in adults at steady state. The study will be conducted in pediatric OAB patients to establish the single-dose PK and the acute safety profile of solifenacin aqueous suspension. Each of the six groups will consist of at least six patients.

The study will start with the lowest dose group in adolescent patients (12 to 17 years). When this group has completed the study, their safety and concentration data will be reviewed by a Safety Review Committee. If no safety concerns are evident according to pre-specified criteria, enrollment of children (5 to 11 years) in the lowest dose group and adolescents in the intermediate dose group will be started simultaneously. When these groups have completed the study, their safety data and drug concentration data will also be reviewed. If no safety concerns occurred, enrollment of children in the intermediate dose group and of adolescents in the highest dose group will be started simultaneously. Finally, after these groups completed the study and no safety concerns occurred during associated data review, enrollment of children in the highest dose group will start. Interim review of plasma exposure at lower doses will be used to adjust the next higher doses administered, if necessary.

ELIGIBILITY:
Inclusion Criteria:

* Symptoms of urgency, diagnosed as OAB according to International Children's Continence Society (ICCS) criteria
* Daytime urgency incontinence at least once/day

Exclusion Criteria:

* Daytime voiding frequency less than 5
* Uroflow indicative of pathology other than OAB
* Maximum voided volume > age expected capacity ([age +1] x 30) in ml
* Post voiding residual (PVR) > 10% of the functional bladder capacity
* Monosymptomatic enuresis
* Congenital anomalies of the genito-urinary tract or nervous system
* Current constipation (when treated the patient can enter the study)
* Current urinary tract infection (patient will be eligible for enrolment 14 days after a negative dipstick test, provided a second dipstick test, performed after these 14 days, is also negative)
* Serum creatinine more than or equal to 2 times the upper limit of normal (ULN)
* Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) more than or equal to 2 times ULN, or bilirubin more than or equal to 1.5 times ULN

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 42 (Actual)
Dates: Start 2010-10-20 (Actual); Primary Completion 2011-08-14 (Actual); Study Completion 2011-08-14 (Actual)

PRIMARY OUTCOMES:
Maximum Concentration (Cmax) | Day 1 predose up to Day 7 postdose
Area Under the Concentration-time Curve Extrapolated to Infinity (AUCinf) | Day 1 predose up to Day 7 postdose
Apparent Terminal Elimination Half-life (t1/2) | Day 1 predose up to Day 7 postdose
Time to Attain Cmax (tmax) | Day 1 predose up to Day 7 postdose
Area Under the Concentration-time Curve from the Time of Dosing Until the Last Measurable Concentration (AUClast) | Day 1 predose up to Day 7 postdose
Apparent Total Body Clearance (CL/F) | Day 1 predose up to Day 7 postdose
Apparent Volume of Distribution During the Terminal Phase (Vz/F) | Day 1 predose up to Day 7 postdose

SECONDARY OUTCOMES:
Number of Participants with Adverse Events (AEs) | From the first dose of study drug up to 7 days postdose
  Safety is monitored by collecting AEs, which includes abnormal laboratory tests, vital signs or ECG data that are defined as an AE if the abnormality induces clinical signs or symptoms, requires active intervention, interruption or discontinuation of study medication or is clinically significant in the investigator's opinion. A treatment-emergent adverse event (TEAE) is defined as an AE that occurs or worsens after study drug administration. A serious AE (SAE) is any untoward medical occurrence that, at any dose: Results in death, is life-threatening, results in persistent or significant disability/incapacity, results in congenital anomaly, or birth defect, requires inpatient hospitalization or leads to prolongation of hospitalization or other medically important events.
Change from baseline in postvoid residual (PVR) volume | Baseline (screening) and 4 hours postdose
  PVR volume is assessed by ultrasonography or bladder scan.

CONTACTS AND LOCATIONS:
Overall Officials: Use Central Contact, Study Chair — Astellas Pharma Europe B.V.
Locations (8):
- Belgium (2):
  - Ghent
  - Kortrijk
- Aarhus, Denmark
- Sweden (2):
  - Gothenburg
  - Uppsala
- United Kingdom (3):
  - Cambridge
  - Manchester
  - Sheffield

IPD SHARING:
Plan to Share IPD: No
Access to anonymized individual participant level data will not be provided for this trial. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.

REFERENCES:
- See also: Link to results on the Astellas Clinical Study Results website — https://astellasclinicalstudyresults.com/study.aspx?ID=243